CLINICAL TRIAL: NCT00333268
Title: Clinical Evaluation of the Safety and Efficacy of Next Generation Ophthalmic Irrigating Solution Compared to BSS Plus for Use During Cataract Extraction and IOL Implantation
Brief Title: Safety and Efficacy of Next Generation Ophthalmic Irrigating Solution Compared to BSS Plus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-04-14
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — glutathione-bicarbonate-Ringer solution

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- NGOIS (Experimental)
  Interventions: Drug: Next Generation Ophthalmic Irrigating Solution (NGOIS)
- BSS Plus (Active Comparator)
  Interventions: Drug: BSS Plus

INTERVENTIONS:
Drug: Next Generation Ophthalmic Irrigating Solution (NGOIS) — Volume sufficient to irrigate adequately during cataract surgery
  Arms: NGOIS
Drug: BSS Plus — Volume sufficient to irrigate adequately during cataract surgery
  Arms: BSS Plus

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Next Generation Ophthalmic Irrigating Solution (NGOIS) compared to BSS Plus for use during cataract extraction and intra-ocular lens (IOL) implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients any race or sex 18 or older and undergoing cataract extraction with planned implantation of a posterior chamber intraocular lens.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Under 18
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2004-09; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Percent change in endothelial cell density

SECONDARY OUTCOMES:
Best corrected logMAR visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- United States, Fort Worth, Texas, United States